CLINICAL TRIAL: NCT06994910
Title: Investigation Into the Effectiveness of Maitland Joint Mobilization in Alleviating Symptoms of Temporomandibular Disorders, Enhancing Joint Function, and Oral Behaviors
Brief Title: Temporomandibular Disorders Physiotherapy
Acronym: TMD/VAS/ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Polytechnic University (Other)
Responsible Party: Principal Investigator, Mohammad Al-Talahma, Assistant Professor, Palestine Polytechnic University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAMS/PTBR/3/127
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular Disorders; Physiotherapy; Maitland Mobilization Technique
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: A single group of participants received the intervention. Outcomes were measured before and after the intervention within the same group to assess changes over time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before Maitland joint mobilization (Experimental): Participants with temporomandibular joint dysfunction received Maitland mobilization techniques applied to the TMJ over a defined treatment period. Outcomes were assessed at baseline (pre-intervention) and after completion of the intervention (post-intervention)
  Interventions: Other: Maitland mobilization techniques
- After Maitland joint mobilization (Experimental): Participants with temporomandibular joint dysfunction received Maitland mobilization techniques applied to the TMJ over a defined treatment period. Outcomes were assessed at baseline (pre-intervention) and after completion of the intervention (post-intervention).
  Interventions: Other: Maitland mobilization techniques

INTERVENTIONS:
Other: Maitland mobilization techniques — Participants with temporomandibular joint dysfunction received Maitland mobilization techniques applied to the TMJ over a defined treatment period. Outcomes were assessed at baseline (pre-intervention) and after completion of the intervention (post-intervention)

SUMMARY:
This study aims to investigate the effectiveness of the Maitland joint mobilization technique in alleviating symptoms related to (temporomandibular disorders) TMD and to investigate its influence on patient clinical outcomes, including pain intensity, TMJ range of motion (ROM), functional limitations, disability, and oral behaviors.

DETAILED DESCRIPTION:
Physiotherapeutic procedures for TMD aim to reduce pain, enhance neuromuscular coordination and strength, and promote joint range of motion (ROM), mastication, mouth opening, and general mobility. The literature highlights a variety of physiotherapy techniques used to treat TMD, including manual therapy, stretching, active and passive exercises, as well as modalities like thermotherapy, ultrasound, electrotherapy, iontophoresis, laser therapy, shockwave therapy, infrared therapy, kinesiology taping, and dry needling. Clinical research supports the efficacy of physiotherapy as a conservative treatment for TMD, effectively addressing pain, muscular dysfunctions, and psychosocial factors. Optimal results are achieved through a combination of therapeutic exercises and manual therapy, which is considered one of the most effective approaches.

The Maitland joint mobilization technique is a key physiotherapeutic procedure for managing TMD. This technique involves passive, rhythmic joint mobilizations aimed at restoring joint functionality and alleviating pain. The technique employs five grades of mobility, each designed for specific therapeutic goals. Grades I and II are used to reduce pain and relax soft tissues, while Grades III, IV, and V focus on addressing joint hypomobility by stretching soft tissues and improving joint mobility. The technique enhances both osteokinematic and arthrokinematic movements, with osteokinematic referring to voluntary joint motion, and arthrokinematic to the small, involuntary movements that occur during normal joint ROM. Maitland joint mobilization utilizes controlled forces in specific directions, based on Kaltenborn's concave-convex rule, to optimize both movements and improve joint function. This research is essential for providing further evidence that supports enhanced physiotherapeutic techniques, resulting in enhancing patient clinical outcomes and enhancing professional practices for the optimal management of TMD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: individuals diagnosed with TMD, whether it is unilateral or bilateral.
* Myofascial pain and myo-spasm.
* Anterior disk displacement with reduction and anterior disk displacement without reduction.
* Craniofacial and craniomandibular pain.
* Myofascial pain with or without limited mouth opening.

Exclusion Criteria:

* Patients with a documented history of surgical procedures involving the TMJ.
* Patients with a confirmed diagnosis of systemic diseases (e.g., rheumatic and metabolic diseases).
* Patients with congenital or developmental craniofacial anomalies, including conditions like as ankylosis.
* Patients with diagnosed cancer.
* Patients with mental, physical disorders and language difficulties.
* Patients with diagnosed neuropathic and dental pain.
* Patients with diagnosed general myopathy (e.g., fibromyalgia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Pain will be measured at baseline (pre-intervention) and after completion of the 4-week intervention (post-intervention)
  Pain intensity will be assessed using a 10-centimeter Visual Analogue Scale (VAS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Participants will be asked to indicate the average intensity of their jaw-related pain experienced over the past week. This tool is used to evaluate the effect of the intervention on subjective pain levels in patients diagnosed with temporomandibular disorders.
Temporomandibular joint range of motion | Temporomandibular joint range of motion will be assessed at baseline (pre-intervention) and after the 4-week intervention (post-intervention).
  The range of motion (ROM) of the temporomandibular joint will be measured using the TheraBiteⓇ Range of Motion Scales, a standardized tool designed to accurately assess mandibular movements including maximum mouth opening, lateral excursion, and protrusion. Measurements will be taken in millimeters by trained assessors to evaluate functional improvement following the intervention in patients with temporomandibular disorders.
Jaw functional disability | Jaw functional disability will be assessed at baseline (pre-intervention) and after the 4-week intervention (post-intervention).
  Jaw functional disability will be evaluated using the Jaw Functional Limitation Scale (JFLS-20), a validated and reliable questionnaire designed to assess limitations in jaw function across three domains: mastication, jaw movements, and verbal communication. Patients will self-report the degree of difficulty experienced during specific functional activities related to the temporomandibular joint. This measure will assess the impact of the intervention on improving jaw function in patients with temporomandibular disorders.
Oral behaviors | Oral behaviors will be assessed at baseline (pre-intervention) and after the 4-week intervention (post-intervention).
  Oral behaviors will be evaluated using the Oral Behavior Checklist (OBC), a validated self-report questionnaire designed to assess the frequency and type of oral behaviors during waking hours and sleep. This includes activities such as clenching, grinding, and other parafunctional habits that may influence temporomandibular disorder symptoms. The OBC will help determine changes in oral behaviors as a result of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Palestine Polytechnic University, Hebron, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after publication of the main results, for a period of 3 years
Access Criteria: IPD and supporting documents (such as the study protocol and statistical analysis plan) will be made available to qualified researchers upon reasonable request. Requests must include a clear research purpose and be approved by an independent ethics committee or institutional review board. Requests can be submitted by email to Dr. Mohammad Al-Talahma at [mtalahma@ppu.edu], and approved data will be shared via secure electronic transfer.

REFERENCES:
- See also: Related Info — https://doi.org/10.1186/s12903-024-03983-7